CLINICAL TRIAL: NCT01382134
Title: Effect of Aspirin, in Vitro Hemodilution and Desmopressin on Platelet Dysfunction Associated With Mild Hypothermia in Healthy Volunteers
Brief Title: Effect of Aspirin, Hemodilution and Desmopressin on Platelet Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tsui Pui Yee, Dr TSUI Pui Yee, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 11-075
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Platelet Dysfunction; Hemodilution; Mild Hypothermia; NSAID; Desmopressin
Keywords: Platelet dysfunction; Hemodilution; Mild hypothermia; NSAID; Desmopressin
MeSH Terms: interventions — Aspirin; Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator): Subjects will be given placebo daily for 3 days. On day 4 an early morning urine sample will be collected for detection of aspirin metabolite (11-dehydro thromboxane B2). On day 6 venous blood sample will be collected, 17mls before and 17 mls after injection of DDAVP 15 microgram subcutaneously. The blood samples will then be subjected for platelet function analysis.
  Interventions: Drug: Placebo, desmopressin
- Aspirin group (Active Comparator): Subjects will be given aspirin 100mg daily for 3 days. On day 4 an early morning urine sample will be collected for detection of aspirin metabolite (11-dehydro thromboxane B2). On day 6 venous blood sample will be collected, 17mls before and 17 mls after injection of DDAVP 15microgram subcutaneously. The blood samples will then be subjected for platelet function analysis.
  Interventions: Drug: Aspirin, desmopressin

INTERVENTIONS:
Drug: Aspirin, desmopressin — Aspirin 100mg daily for 3 days Desmopressin 15 microgram subcutaneously once only
  Arms: Aspirin group
Drug: Placebo, desmopressin — Placebo 1 tab daily for 3 days Desmopressin 15 microgram subcutaneously once only
  Arms: Placebo group

SUMMARY:
Study hypothesis: Desmopressin (DDAVP) can improve platelet function under influence of aspirin, hemodilution and mild hypothermia

Mild hypothermia (34-35oC) is known to cause platelet dysfunction. This could lead to increased surgical bleeding and increased transfusion requirement during surgery. Although this hypothermia-induced platelet dysfunction seems to be reversible with warming, this is not always possible or desirable.

Desmopressin (DDAVP) is a drug which has proven efficacy in improving platelet function in uraemic and cirrhosis patients, and in reducing blood loss in selected surgeries. In a recent study, we have found that subcutaneous injection of 1.5 mcg (1/10th the usual dose) is already sufficient to fully reverse the platelet dysfunction seen at 32oC. We have demonstrated in another study that prolongation of the bleeding time in a 20% hemodiluted sample predicts increased postoperative bleeding after total knee replacement.

We have therefore designed this study as a follow up to our last two studies on DDAVP and hypothermia, to investigate whether hemodilution affects hypothermia induced platelet dysfunction and the response to DDAVP. In addition, another common cause of perioperative platelet dysfunction is the intake of COX inhibitors, particularly aspirin by patients. Therefor the effect of aspirin on hypothermia induced platelet dysfunction and the response to DDAVP, will also be investigated.

DETAILED DESCRIPTION:
Mild hypothermia (34-35oC) is known to cause platelet dysfunction. Increased surgical bleeding and increased transfusion requirement at this temperature range has been reported in both cardiac and noncardiac surgeries. This degree of hypothermia is common during any general anaesthesia, particularly during surgeries which invlove major fluid shift and large area exposure of patients, e.g. trauma and burn patients.

Although this hypothermia-induced platelet dysfunction seems to be reversible with warming, warming is not always possible or desirable. During major trauma or burn surgery, surface warming of patient is practically difficult. During surgeries with major blood loss and fluid shift, heat loss usually occurs at a rate that is more rapid than any warming device can catch up with. During neurosurgery, cooling may be beneficial to neurological outcome.

Desmopressin (DDAVP) is a drug which has proven efficacy in improving platelet function in uraemic and cirrhosis patients, and in reducing blood loss in selected surgeries. In a previous in vitro study, we have found that desmopressin significantly improves platelet function at 32oC. The improvement is seen with a very low concentration of desmopressin in vitro, which suggests that probably doses much smaller than the "standard dose" (15 mcg slow iv or subcutaneous) may be useful. In keeping with this in vitro study, in a more recent study, we have found that subcutaneous injection of 1.5 mcg (1/10th the usual dose) is already sufficient to fully reverse the platelet dysfunction seen at 32oC.

One of the limitations of our previous two studies is that the degree of platelet dysfuction observed at 32oC is relatively mild, with only around 20% prolongation of the closure times on the PFA-100® platelet function analyser. The clinical significance of such prolongation remains uncertain. However, we have demonstrated previously in another study that prolongation of the closure time to >188 sec in a 20% hemodiluted sample predicts increased postoperative bleeding after total knee replacement. We have therefore designed this study as a follow up to our last two studies on DDAVP and hypothermia, to investigate whether hemodilution affects hypothermia induced platelet dysfunction and the response to DDAVP.

In addition, another common cause of perioperative platelet dysfunction is the intake of COX inhibitors, particularly aspirin by patients. Therefor the effect of aspirin on hypothermia induced platelet dysfunction and the response to DDAVP, will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* 60 adult Chinese subjects aged 18-60 without known platelet disorder, thrombocytopenia, history of taking drugs that may affect platelet function including herbal preparations.

Exclusion Criteria:

1. Any known platelet or coagulation disorder
2. Expected surgical operation or dental treatment within one week of scheduled drug intake.
3. Known peptic ulcer disease
4. Obesity (BMI >=30)
5. Pregnant or lactating women.
6. Known chronic liver or renal disease.
7. Coronary artery, carotid artery or peripheral artery disease
8. Recent history of taking antiplatelet drugs, anticoagulants or herbal preparations.
9. Smoker or alcohol user
10. Mentally incapable of providing informed consent
11. Students or junior staff members who had direct working relationship with the PI

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Platelet function | Day 6 after aspirin intake
  Venous blood sample will be taken from subjects before and after injection of DDAVP. Blood sample will be subjected to: (i) complete blood count, (ii) PFA-100 platelet function analyzer, (iii) fibrinogen, and (iv) vWF:Ag concentration for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, China

REFERENCES:
- [Background] Wolberg AS, Meng ZH, Monroe DM 3rd, Hoffman M. A systematic evaluation of the effect of temperature on coagulation enzyme activity and platelet function. J Trauma. 2004 Jun;56(6):1221-8. doi: 10.1097/01.ta.0000064328.97941.fc. PMID 15211129
- [Background] Cavallini M, Baruffaldi Preis FW, Casati A. Effects of mild hypothermia on blood coagulation in patients undergoing elective plastic surgery. Plast Reconstr Surg. 2005 Jul;116(1):316-21; discussion 322-3. doi: 10.1097/01.prs.0000170798.45679.7a. PMID 15988284
- [Background] Michelson AD, Barnard MR, Khuri SF, Rohrer MJ, MacGregor H, Valeri CR. The effects of aspirin and hypothermia on platelet function in vivo. Br J Haematol. 1999 Jan;104(1):64-8. doi: 10.1046/j.1365-2141.1999.01146.x. PMID 10027713
- [Background] Hofer CK, Worn M, Tavakoli R, Sander L, Maloigne M, Klaghofer R, Zollinger A. Influence of body core temperature on blood loss and transfusion requirements during off-pump coronary artery bypass grafting: a comparison of 3 warming systems. J Thorac Cardiovasc Surg. 2005 Apr;129(4):838-43. doi: 10.1016/j.jtcvs.2004.07.002. PMID 15821652
- [Background] Schmied H, Kurz A, Sessler DI, Kozek S, Reiter A. Mild hypothermia increases blood loss and transfusion requirements during total hip arthroplasty. Lancet. 1996 Feb 3;347(8997):289-92. doi: 10.1016/s0140-6736(96)90466-3. PMID 8569362
- [Background] Winkler M, Akca O, Birkenberg B, Hetz H, Scheck T, Arkilic CF, Kabon B, Marker E, Grubl A, Czepan R, Greher M, Goll V, Gottsauner-Wolf F, Kurz A, Sessler DI. Aggressive warming reduces blood loss during hip arthroplasty. Anesth Analg. 2000 Oct;91(4):978-84. doi: 10.1097/00000539-200010000-00039. PMID 11004060
- [Background] Schmied H, Schiferer A, Sessler DI, Meznik C. The effects of red-cell scavenging, hemodilution, and active warming on allogenic blood requirements in patients undergoing hip or knee arthroplasty. Anesth Analg. 1998 Feb;86(2):387-91. doi: 10.1097/00000539-199802000-00032. PMID 9459254
- [Background] Todd MM, Hindman BJ, Clarke WR, Torner JC; Intraoperative Hypothermia for Aneurysm Surgery Trial (IHAST) Investigators. Mild intraoperative hypothermia during surgery for intracranial aneurysm. N Engl J Med. 2005 Jan 13;352(2):135-45. doi: 10.1056/NEJMoa040975. PMID 15647576
- [Background] Ying CL, Tsang SF, Ng KF. The potential use of desmopressin to correct hypothermia-induced impairment of primary haemostasis--an in vitro study using PFA-100. Resuscitation. 2008 Jan;76(1):129-33. doi: 10.1016/j.resuscitation.2007.07.009. Epub 2007 Aug 21. PMID 17714852
- [Background] Ng KF, Lawmin JC, Tsang SF, Tang WM, Chiu KY. Value of a single preoperative PFA-100 measurement in assessing the risk of bleeding in patients taking cyclooxygenase inhibitors and undergoing total knee replacement. Br J Anaesth. 2009 Jun;102(6):779-84. doi: 10.1093/bja/aep091. Epub 2009 May 2. PMID 19411670
- [Background] Gallinaro L, Cattini MG, Sztukowska M, Padrini R, Sartorello F, Pontara E, Bertomoro A, Daidone V, Pagnan A, Casonato A. A shorter von Willebrand factor survival in O blood group subjects explains how ABO determinants influence plasma von Willebrand factor. Blood. 2008 Apr 1;111(7):3540-5. doi: 10.1182/blood-2007-11-122945. Epub 2008 Feb 1. PMID 18245665
- [Background] Mannucci PM, Capoferri C, Canciani MT. Plasma levels of von Willebrand factor regulate ADAMTS-13, its major cleaving protease. Br J Haematol. 2004 Jul;126(2):213-8. doi: 10.1111/j.1365-2141.2004.05009.x. PMID 15238142
- [Derived] Tsui PY, Cheung CW, Lee Y, Leung SW, Ng KF. The effectiveness of low-dose desmopressin in improving hypothermia-induced impairment of primary haemostasis under influence of aspirin - a randomized controlled trial. BMC Anesthesiol. 2015 May 28;15:80. doi: 10.1186/s12871-015-0061-5. PMID 26017715